CLINICAL TRIAL: NCT07107334
Title: A Pilot Study to Estimate Early Clinical Efficacy Signals of a Glucagon-like Peptide 1 Receptor Agonist (GLP-1RA) Administration in Conjunction With Levonorgestrel Intrauterine Device (LNG-IUD) in Obese Patients With Endometrioid Intraepithelial Neoplasia
Brief Title: A Study to Estimate Early Clinical Efficacy Signals of GLP-1 Agonist Administration in Conjunction With Levonorgestrel Intrauterine Device in Obese Patients With Endometrioid Intraepithelial Neoplasia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF-GYN-XXX
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Endometrioid Endometrial Adenocarcinoma
Keywords: Endometrial cancer; endometrial intraepithelial neoplasia; endometrial adenocarcinoma; Levonorgestrel IUD
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glucagon-like peptide 1 receptor agonist (Experimental)
  Interventions: Drug: Glucagon-like peptide 1 receptor agonist

INTERVENTIONS:
Drug: Glucagon-like peptide 1 receptor agonist — Subjects will receive a glucagon-like peptide 1 receptor agonist by self-injection for as long as clinically indicated by the treating physician or until the subject receives clearance for staging hysterectomy or for pregnancy pursuit. The choice of glucagon-like peptide 1 receptor agonist for each subject will be at the treating physician's discretion. Subjects will discontinue the glucagon-like peptide 1 receptor agonist 2 weeks before any elective surgical procedure.

SUMMARY:
This study will explore the use of glucagon-like peptide 1 receptor agonist (GLP-1RA) used concurrently with levonorgestrel intrauterine device in patients with poor surgical candidacy for a hysterectomy or patients who are pursuing fertility sparing. GLP-1RA are a class of medications that mimic the natural hormone glucagon-like peptide-1. These medications trigger the pancreas to release insulin which can help lower blood sugar levels and delay gastric emptying. The recent FDA approval of GLP-1RAs has changed the landscape for pharmacotherapy for weight loss. These hormone-based obesity medications are novel and revolutionary in obesity medicine. Liraglutine, semaglutide, and tirzepatide have become exceedingly popular for their effects on weight loss and obesity-related comorbidities. More recently, GLP-1RAs have exhibited risk reduction of various obesity associated cancers, including endometrial cancer but their exact role in prevention and treatment has yet to be measured.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* A pathological diagnosis with in the past 3 months consistent with grade 1 endometrioid endometrial adenocarcinoma or endometrial intraepithelial neoplasia
* ECOG Performance Status of 0 to 3
* No extrauterine involvement or myometrial invasion by MRI (preferred) or transvaginal ultrasound with in the last 3 months
* BMI ≥ 30 kg/m2 and one of the following:

  1. Multiple medical co-morbidities (defined as American Society of Anesthesiologists [ASA] score ≥ 3) at physician discretion
  2. Fertility desire
* Subjects must not have more than one active malignancy at the time of enrollment (Subjects with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the study [as determined by the treating physician or approved by the Principal Investigator] may be included).
* Written informed consent obtained from the subject and the subject agrees to comply with all the study-related procedures.

Exclusion Criteria:

* Subjects with grade 2 or 3 endometroid or any non-endometrioid histology (i.e., clear cell, carcinoma, serous)
* Subjects whose tumors are estrogen receptor negative
* Clinical suspicion of metastatic disease as assessed by the treating physician or confirmed metastatic disease based on imaging
* Subjects with abnormal cervical cytology
* Subjects who are diagnosed with thyroid cancer, pancreatitis, or multiple endocrine neoplasia syndrome type 2
* Subjects who are confirmed to be pregnant or breastfeeding
* History of medullary thyroid cancer
* History of any other disease, metabolic dysfunction, clinical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of protocol therapy or that might affect the interpretation of the results of the study or that puts the subject at high risk for treatment complications, in the opinion of the treating physician.
* Prisoners or subjects who are involuntarily incarcerated, or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Time from start of GLP-1RA to clearance of staging hysterectomy | 12 months
  Determine the time from start of GLP-1RA treatment to clearance for staging hysterectomy in patients with poor surgical candidacy for a hysterectomy.
Time from start of GLP-1RA to clearance for pregnancy pursuit | 12 months
  Determine the time from start of GLP-1RA treatment to clearance for pregnancy pursuit in patients pursuing fertility sparing.
Endometrial pathologic response | 6 months after beginning GLP-1RA treatment
  Determine the endometrial pathologic response 6 months after beginning GLP-1RA treatment
Endometrial pathologic response | 12 months after beginning GLP-1RA treatment
  Determine the endometrial pathologic response 12 months after beginning GLP-1RA treatment

SECONDARY OUTCOMES:
Length of surgery | Intraoperative
  Determine the length of staging hysterectomy surgery
Number of nights in hospital | 12 months
  Determine the number of nights spent in the hospital for staging hysterectomy
Postoperative complications | 12 months
  Determine the postoperative complications following staging hysterectomy
Patient-reported quality of life | 6 months
  Compare patient-reported quality of life, as measured by the EORTC QLQ-C30, v3.0 between baseline and at 6 months after beginning GLP-1RA treatment
Patient-reported quality of life | 12 months
  Compare patient-reported quality of life, as measured by the EORTC QLQ-C30, v3.0 between baseline and at 12 months after beginning GLP-1RA treatment
Patient-reported quality of life | at either clearance for pregnancy pursuit or staging hysterectomy, which will ideally occur by 12 months after beginning study treatment
  Compare patient-reported quality of life, as measured by the EORTC QLQ-C30, v3.0 between baseline and at end of GLP-1RA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kaitlin Nicholson, MD, Principal Investigator — University of Florida